CLINICAL TRIAL: NCT01655758
Title: The 24 Control of IOP in Ocular Hypertension: a Cross-over Study on Inflow Versus Outflow Drugs.
Brief Title: 24-hour Control of Intraocular Pressure (IOP) in Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Stefano Gandolfi, professor of ophthalmology and chairman,, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UParma2004crossover
Record Dates: First submitted 2012-07-21; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Ocular Hypertension
Keywords: glaucoma; 24-hour IOP; outflow drugs; inflow drugs
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Timolol; dorzolamide-timolol combination; Latanoprost; Travoprost; methylacetylene; Bimatoprost

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- timolol (Active Comparator): 60-day treatment phase with 0.5% timolol eyedrops, b.i.d.
  Interventions: Drug: 0.5% timolol
- 'timolol-dorzolamide fixed combination' (Active Comparator): 60-day treatment phase with the fixed combination of 0.5% timolol-2% dorzolamide, eyedrops, b.i.d.
  Interventions: Drug: timolol-dorzolamide fixed combination
- xalatan (Active Comparator): 60-day treatment phase with 0.005% latanoprost, eyedrops, QD
  Interventions: Drug: Latanoprost
- travatan (Active Comparator): 60-day treatment phase with 0.004% travoprost, eyedrops, QD
  Interventions: Drug: Travoprost
- lumigan (Active Comparator): 60-day treatment phase with 0.03% bimatoprost, eyedrops, QD
  Interventions: Drug: Bimatoprost

INTERVENTIONS:
Drug: 0.5% timolol
  Other Names: timoptol (MSD)
  Arms: timolol
Drug: timolol-dorzolamide fixed combination
  Other Names: cosopt (MSD)
  Arms: 'timolol-dorzolamide fixed combination'
Drug: Latanoprost
  Other Names: xalatan (pfizer)
  Arms: xalatan
Drug: Travoprost
  Other Names: travatan (Alcon)
  Arms: travatan
Drug: Bimatoprost
  Other Names: lumigan (Allergan)
  Arms: lumigan

SUMMARY:
This study was designed to compare the 24-hour efficacy on intra ocular pressure (IOP) of drugs acting either on aqueous humor production ("inflow drugs") or on aqueous humor outflow ("outflow drugs") in human eyes affected by ocular hypertension and virgin to treatment. The enrolled patients will be exposed, in a cross-over design, to n = 2 aqueous suppressants and n= 3 uveoscleral outflow enhancers, and 24 hr IOP will be measured. It is hypothesised that outflow drugs may offer a better and more stable control of IOP through the 24 hours.

DETAILED DESCRIPTION:
(a) study design: Prospective, open label, investigator-masked clinical trial, with cross-over design, both eyes treated, OD chosen for analysis; (b) study population: patients, showing ocular hypertension, who were never exposed to hypotensive treatment (see inclusion and exclusion criteria for details). (c) study drugs: Timolol and dorzolamide will be chosen as inflow drugs. The three prostaglandin analogues (PGA) Latanoprost, travoprost and bimatoprost will be chosen as outflow drugs. (d) study flow-chart: upon enrollment, patients will be initiated to the following schedule: 60 days timolol 0.5% bid, 60 days washout, 60 days timolol 0.5%-dorzolamide 2% fixed combination bid, 60 days washout, 60 days PGA1, 60 days washout, 60 days PGA2, 60 days washout, 60 days PGA3. Patients were assigned to the PGAs according to a sequence (L-T-B) randomly generated. Data will be collected at baseline and at the and of each study phase (i.e. active treatment and washout)(e) main efficacy outcome: change in the mean IOP (with respect to baseline) at the end of each study phase and change of IOP (with respect to baseline) at the different time points of the 24-hour phasing. IOP will be measured at 8 a.m., 11 a.m., 3 p.m., 6 p.m. and 9 p.m. by means of Goldmann applanation tonometry at the slit lamp. At midnight, 2 a.m. and 6 a.m. the Tonopen in supine position will be used. (f) statistics: the analysis of co-variance (ANCOVA) for paired samples with Bonferroni correction will be adopted. A minimum sample size of 51 patients is needed for a minimal expected difference in mean IOP between inflow and outflow drugs = 2.5 mmHg, with an estimated pooled variance = 4 , a power = 90% and an alpha probability = 5%.

ELIGIBILITY:
Inclusion Criteria:

* IOP > 22 mmHg and < 30 mmHg on at least three readings on separate days ,
* Open angle on gonioscopy,
* CCT > 550 m,
* optic disk classified as "within normal limits" by Moorfields Regression analysis, HRTII,
* normal visual field (standard achromatic perimetry, Humphrey Field Analyzer, 24/2 SITA standard),
* Age > 40 and < 70 years,
* refraction between - 5 and + 2 dyopters,
* best corrected visual acuity better than 0.2 LogMAR,

Exclusion Criteria:

* PEX
* PDS
* ocular comorbidiities other than refractive problems and/or mild dry eye
* history of diabetes
* treatment with systemic beta blockers and steroids
* previous treatment with ocular hypotensive drugs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-01; Primary Completion 2003-12 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
change in the mean IOP at the end of each phase vs baseline, and change of IOP at the different time points of the 24-hour phasing with respect to baseline | IOP will be measured, at baseline, on day 60, 120, 180, 240, 300, 360,420,480 and 540, at 8 a.m., 11 a.m., 3 p.m., 6 p.m., 9 p.m., midnight, 2 a.m. and 6 a.m.
  Goldmann Applanation tonometry (GAT): 2 readings averaged. If >2 mmHg difference between the two, a further reading will be performed. GAT will be adopted during the day, and performed at the slit lamp in sitting position.
  Tonopen: 4 readings averaged. Tonopen will be used during the night, and the measurements will be perfomred on patients laying in bed in supine position.

SECONDARY OUTCOMES:
visual field | visual field (24/2 SITA) will be performed at screening and at the end of the study (i.e. upon completion of the last cross-over arm, 540 days after baseline)
  Humphrey Field Analyzer, 24/2 SITA standard

CONTACTS AND LOCATIONS:
Overall Officials: STEFANO GANDOLFI, MD, Principal Investigator — University of Parma
Locations (1):
- University Eye Clinic, Parma, Italy